CLINICAL TRIAL: NCT04537858
Title: Analysis of the Influence of Rehabilitation With Virtual Reality on the Heart Rate Variability of Individuals Under Treatment of COVID-19 in a Hospital Unit.
Brief Title: Virtual Reality Therapy Influence on Heart Rate Variability of Inpatients With COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Talita Dias da Silva, Researcher, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 33244620.5.0000.5505
Record Dates: First submitted 2020-08-29; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: COVID-19; Inpatient
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality therapy first (Experimental): Subjects with COVID-19 who will start the first day of the protocol with Virtual Reality tasks in the morning and then in the second period, in the afternoon, will perform the conventional exercises (n = 25)
  Interventions: Device: Virtual reality therapy first
- Conventional therapy first (Experimental): Subjects with COVID-19 who will start the first day with conventional exercises in the morning and in the second period, in the afternoon, will perform activity with virtual reality (n = 25).
  Interventions: Device: Conventional therapy first

INTERVENTIONS:
Device: Virtual reality therapy first — First day of the protocol with Virtual Reality intervention in the morning and conventional intervention in the afternoon
  Arms: Virtual reality therapy first
Device: Conventional therapy first — First day of the protocol with conventional intervention in the morning and Virtual Reality intervention in the afternoon
  Arms: Conventional therapy first

SUMMARY:
The end of 2019 saw the emergence of a new human coronavirus (COVID-19) spread rapidly around the world and has a high degree of lethality. In more severe cases, patients remain in hospital inpatient units, under the care of the health team. To serve this population, it is important to use and develop potential tools to meet the demands of physical activity and improve cardiorespiratory fitness. In this sense, exposure therapies of virtual reality are promising and, although limited for this purpose, have been shown to be an adequate and equivalent alternative to traditional exercise programs. Fifty patients with confirmed diagnosis of COVID-19 will be evaluated in an inpatient unit at Hospital São Paulo, at Escola Paulista de Medicina, Universidade Federal de São Paulo (HSP - EPM/UNIFESP). After completing all the questionnaires and tests of the initial evaluation (Medical Research Council Scale, Visual Analogue Scale, BORG Scale, Brunel's Mood Scale, Satisfaction Scale and Heart Rate Variability - HRV), the individuals will be divided into two groups being Group A: Subjects with COVID-19 who will start the first day of the protocol with Virtual Reality tasks in the morning and then in the second period, in the afternoon, will perform the conventional exercises (n = 25); And Group B: Subjects with COVID-19 who will start the first day with conventional exercises in the morning and in the second period, in the afternoon, will perform activity with virtual reality (n = 25). After the application of therapies, final evaluations will be carried out. The rehabilitation protocol will be applied during all days of hospitalization. For the protocol, the Heart Rate Variability indices will be evaluated in three moments: (1) rest before the task, (2) during the intervention, (3) recovering from the intervention. The performance data during the activity in Virtual reality will also be evaluated. The results of this study will assist in assessing the response to rehabilitation therapies during hospitalization and the prognosis of these patients.

DETAILED DESCRIPTION:
To carry out this study, an experimental protocol will be used, where patients admitted to an inpatient unit of the São Paulo hospital will perform a rehabilitation protocol at two different times using virtual reality tasks and conventional therapies.

In the first moment, in the initial evaluation, only on the first day of care with the patient, the Medical Research Council Scale, Visual Analog Scale, BORG Scale, Brunel Mood Scale and Satisfaction Scale will be applied. At the end of the therapy, a BORG scale is applied to assess and monitor the patient's perception of effort. For the evaluation and characterization of the sample will be used:

Medical Research Council scale (MRC)

The Medical Research Council (MRC) was created in 1943, it is an instrument adapted to assess muscle strength in critically ill patients. The result is obtained through the evaluation of six movements of upper limbs (upper limbs) and lower limbs (lower limbs) and the strength is graded between 0 (plegia) to 5 points (normal strength). The maximum sum can reach 60 points, values below 48 are considered that the patient has muscle weakness.

Visual Analog Scale (EVA) The visual analog scale (VAS) is an instrument to assess the degree of pain in the patient, it consists of a 10 cm line that has, in general, the phrases "absence of pain and unbearable pain" as extremes.

Borg scale

The Borg scale is a tool for monitoring the intensity of physical effort, it is considered as one of the most used instruments for the evaluation and quantification of the sensations of physical effort, also known as subjective perception of effort (PSE). This is used both in the area of high performance sports and in the area of physical rehabilitation, to monitor the changes caused by physical exercise in the cardiorespiratory, metabolic, neuromuscular systems.

Satisfaction Scale (EVA-S)

The 10 cm Visual Analogue Scale (VAS) assesses the level of satisfaction of the interviewed individuals. Patients will answer the questionnaire, and they will be asked to mark with a vertical line at the scale location that indicates satisfaction with rehabilitation, in which zero (0) indicates very dissatisfied and 10 indicates very satisfied.

This scale was developed to allow a quick measurement of the mood of adults and adolescents.

BRUMS contains 24 simple mood indicators, such as feelings of anger, disposition, nervousness and dissatisfaction that are noticeable by the individual being assessed. The evaluated responds the scale according to how they feel about such sensations.

The score is 5 points (0 = nothing to 4 = extremely). The form put in the question is "How do you feel now", although other forms: "How have you felt this past week, including today", or "How do you normally feel" can be used. BRUMS takes about one to two minutes to respond.

The 24 indicators on the scale comprise six subscales: anger, confusion, depression, fatigue, tension and vigor.

Respiratory Rate (RR)

Respiratory rate (RR) is defined as the number of breaths a person takes 1 minute (breaths / min), being an important vital sign. It varies in response to metabolic demand and the normal range for an adult is 12 to 20 breaths.

Before starting therapy with VR and conventional therapy, RF will be measured. At the end of the respective therapies, the RF will be checked again.

Heart Rate (HR)

All heart rate records will be performed using a cardiofrequency meter (V800, Polar). After placing the brace and monitor, individuals will be placed in supine position and will remain at rest breathing spontaneously for 15 minutes and then for another 10 minutes during interventions, whether during VR or conventional.

Oxygen Saturation (Spo2)

Pulse oximetry is widely used for patients who need continuous monitoring of oxygen saturation. Its main purpose is the early detection of hypoxemia in various situations and the monitoring of perfusion and circulation. It is a non-invasive monitoring.

Heart Rate Variability (HRV)

HRV is a simple, reliable, inexpensive and non-invasive measure to capture autonomic impulses. The widespread use and cost-effectiveness of the technique and the ease of data acquisition make HRV a capable choice for the interpretation of cardiac autonomic functioning and a promising clinical tool to assess and identify physiological changes. Fluctuations in HRV patterns provide an early and sensitive diagnosis of the human body's physiological behavior and the individual's health status.

HRV has emerged as a simple and non-invasive measure of autonomic impulses, representing one of the most promising quantitative markers of autonomic balance. HRV describes oscillations in the interval between consecutive heartbeats (R-R intervals), as well as oscillations between consecutive instantaneous heart rates. It is a measure that can be used to assess the modulation of the ANS under physiological conditions, such as in waking and sleeping situations, different body positions, physical training, and also in pathological conditions. Changes in HRV patterns provide a sensitive and early indicator of health impairments

Virtual Reality Training

Participants will perform the tasks individually in a room equipped with a computer, table and chair, in the presence of the evaluator responsible for providing the instructions and recording the results. The chair and footrest will be adjusted according to the individual's height and needs, so that they are positioned correctly during the task. Participants will be instructed to sit in a way they think is most comfortable.

Before starting the task, the researcher will explain the task verbally and will demonstrate how the game works. Then, participants will complete a one-time trial in order to verify that they understand the instructions.

Intervention After performing all the tests and questionnaires of the initial evaluation, individuals will be divided into two groups, being Group A: Subjects with COVID -19 who will start the first day of the protocol with Virtual Reality tasks in the morning and then in the second period in the afternoon, they will perform conventional exercises (n = 25); And Group B: Subjects with COVID -19 who will start the first day with conventional exercises in the morning and in the second period, in the afternoon, will perform activity with virtual reality (n = 25). After the application of therapies, final evaluations will be carried out. The rehabilitation protocol will be applied during hospitalization.

Participants will perform the virtual tasks individually in a room equipped with a computer, table and chair, in the presence of the evaluator responsible for providing the instructions and recording the results. The chair and footrest will be adjusted according to the individual's height and needs, so that they are positioned correctly during the task. Participants will be instructed to sit in a way they think is most comfortable.

Before starting the task, the researcher will explain clearly and objectively how the game works. Then, participants will complete a one-time attempt to make sure they understand the instructions.

MoveHero

Software developed at the School of Arts, Sciences and Humanities of the University of São Paulo will be used. The game features balls that fall, in four imaginary columns on the computer screen, to the rhythm of the chosen music. The task is not to let the balls fall. However, the balls can only be touched when they reach four circles placed in parallel (at two height levels), two on the left and two on the right of the participant (0 0 \ o / 0 0), called targets 1, 2 , 3 and 4, as viewed from left to right.

The game captures the participant's movements through a webcam, not requiring physical contact to perform the task, so the participant must move his arms, at a distance of one and a half meters from the computer screen. The participant must wait for the balls to fall, until they begin to overlap one of the target circles. Therefore, the game requires the participant to have a strategy of anticipating the movement to reach the balls within those circles.

The game offers hit feedback through a numbering (+1) that appears next to the sphere that has been successfully hit within the target, in addition, the total score is visible in the upper left corner of the screen, with 10 points for each hit.

Conventional task

Participants will perform the tasks individually in the inpatient sector, in the presence of the evaluator responsible for providing instructions and recording the results.

Statistical analysis Statistical analyzes will be performed using IBM-SPSS (version 26.0, IBM Corp., Armonk, NY, USA). As dependent variables, all HRV indices will be considered. If the data meet the assumptions of normality, Multiple Analysis of Variances (MANOVA) will be used to compare the study groups (Virtual Group and Conventional Group) and intra-group comparison (virtual and conventional group, when comparing the same subject), with Minimum Significant Difference (LSD) post-test. If the data do not meet the assumptions of normality, the differences between the groups will be analyzed using the Kruskal-Wallis test. Dunn's post hoc tests will be performed on each pair of groups, with Dunn-Bonferroni post-test on each pair of groups66. Values of p <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with confirmed diagnosis of COVID-19.

Exclusion Criteria:

* Cardiac arrhythmias and atrioventricular block,
* Congenital anomalies, such as congenital heart disease,
* Pulmonary malformations,
* Drugs that interfere with SNA, such as anti-arrhythmic drugs.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | 3 months
  Assessment of heart rate variability indices before, during and in the recovering of intervention in order to access autonomic behavior during both interventions and to access behavior of the disease while in the hospital unit.
Motor Skills | 3 months
  Assessment of motor skills, such as improvement in accuracy and precision of movement provided by the games developed for rehabilitation. The variables will be coincident timing evaluation, motor learning variables and performance.

SECONDARY OUTCOMES:
Strength | 3 months
  Strength will be assessed by Medical Research Council Scale, which grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle. The higher the grade, the stronger the muscle.
Perceived Exertion | 3 months
  Perceived Exertion will be assessed through Perceived Exertion Borg Scale. It matches how hard you feel you are working with numbers from 6 to 20, the higher the more you feel.
Satisfaction using the technology | 3 months
  Satisfaction using the technology will be assessed by using Satisfaction Scale. Patients will tick at the scale location that indicates satisfaction with rehabilitation, where zero (0) indicates very dissatisfied and 10 indicates very satisfied.
Mood | 3 months
  Mood will be assessed through BRUMS scale, which contains 24 simple mood indicators, such as feelings of anger, disposition, nervousness and dissatisfaction that are noticeable by the individual being assessed. The evaluated responds the scale according to how they feel about such sensations. The score is 5 points (0 = nothing to 4 = extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Talita D da Silva, Ph.D., Principal Investigator — Universidade Federal de São Paulo
Locations (1):
- Comitê de Ética da Universidade Federal, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] da Silva TD, de Oliveira PM, Dionizio JB, de Santana AP, Bahadori S, Dias ED, Ribeiro CM, Gomes RA, Ferreira M, Ferreira C, de Moraes IAP, Silva DMM, Barnabe V, de Araujo LV, Santana HBR, Monteiro CBM. Comparison Between Conventional Intervention and Non-immersive Virtual Reality in the Rehabilitation of Individuals in an Inpatient Unit for the Treatment of COVID-19: A Study Protocol for a Randomized Controlled Crossover Trial. Front Psychol. 2021 Feb 24;12:622618. doi: 10.3389/fpsyg.2021.622618. eCollection 2021. PMID 33716889